CLINICAL TRIAL: NCT04522869
Title: Evaluation Safety and Efficacy of Umbilical Cord Derived Mesenchymal Stem Cell (UC -MSC) Transplantation for Children Suffering From Liver Cirrhosis Due to Biliary Atresia: A Matched Control Prospective Study
Brief Title: Umbilical Cord Derived Mesenchymal Stem Cell (UC -MSC) Transplantation for Children Suffering From Biliary Atresia
Acronym: UCMSCBA
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Vinmec Research Institute of Stem Cell and Gene Technology (Other)
Collaborators: Number 2 Children's Hospital, Ho Chi Minh City (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ISC.19.10
Record Dates: First submitted 2019-09-04; First posted 2020-08-21 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Primary Biliary Cirrhosis
Keywords: liver cirrhosis; biliary atresia; Kasai's operation
MeSH Terms: conditions — Liver Cirrhosis, Biliary; Liver Cirrhosis; Biliary Atresia | interventions — Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Umbilical cord blood - derived mesenchymal stem cells (Experimental): 17 patients with BA underwent Kasai operation and then will received two doses of UC-MSCs at 1x106 cells/kg (body weight) administered via hepatic artery
  Interventions: Biological: Umbilical Cord Derived Mesenchymal Stem Cell (UC -MSC) Transplantation
- Control group (No Intervention): 17 patients with BA will be conducted Kasai operation only

INTERVENTIONS:
Biological: Umbilical Cord Derived Mesenchymal Stem Cell (UC -MSC) Transplantation — Umbilical Cord Derived Mesenchymal Stem Cell (UC -MSC) Transplantation for Children Suffering From Liver Cirrhosis Due to Biliary Atresia
  Arms: Umbilical cord blood - derived mesenchymal stem cells

SUMMARY:
Biliary atresia (BA) is the most frequent cause of chronic cholestasis in neonates, accounting for at least 50% of pediatric liver transplantation. BA incidence is estimated to range from 1:5000 to 1:19000 live births. All patients will die due to complications of liver cirrhosis if the operation is not performed. Recently, mesenchymal stem cell (MSC) transplantation has been found as a promising therapy for liver cirrhosis in adults. Bone marrow-derived stem cell transplantation was also performed successfully for children with BA. Compared to MSC isolation from bone marrow, isolating MSCs from umbilical cord (UC) tissue is a less invasive procedure.

Furthermore, UC-derived MSCs (UC-MSCs) have been demonstrated to be safe and effective for liver cirrhosis in adults and different pediatric diseases, including liver cirrhosis due to primary biliary cirrhosis. The investigators will compare the outcomes of 17 Kasai operated BA patients who receive UC-MSC transplantation to 17 BA patients who only undergo Kasai operation. Two transplantations of UC - MSCs will be performed via the hepatic artery: the first transplant will be performed at baseline, and the second one will be performed 6 months later with a dosage of 1 million MSCs per kg of body weight. The frequency and severity of the adverse events or serious adverse events associated with UC-MSC injection at 72 hours post-injection will be used to assess the safety. The efficacy of the therapy will be measured using Pediatric End-Stage Liver Disease (PELD) score, liver function, and liver biopsy. This study would open a novel cell therapy to improve outcomes of patients with BA.

DETAILED DESCRIPTION:
The study protocol was approved by the Vinmec International Hospital Ethics Committee, and National Ethics Committees. The stem cell products are conducted in accordance with (GMP) requirements and Good Clinical Practice (GCP). All patients and primary caregivers will receive a written consent form, a cover letter and a clear explanation of the safety issues, potential risks and benefits, and the procedure involved. Moreover, patients will be provided the updated results related to disease and the study during conducting the study and will be fully funded by the project.

ELIGIBILITY:
Inclusion Criteria:

* Children diagnosed with liver cirrhosis due to biliary atresia after Kasai's operation
* From 5 months to 2 years old
* Weight ≥ 6 kg
* Patients with manifestation of cirrhosis on liver biopsy during Kasai's operation.
* Parents or primary caregivers signed the informed consent form.

Exclusion Criteria:

* Under 6kg or over 2 years old
* Coagulation disorders
* Allergy to anesthetic agents
* Active infections

Ages: 5 Months to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2019-08-10 (Actual); Primary Completion 2021-09-25 (Actual); Study Completion 2021-10-25 (Actual)

PRIMARY OUTCOMES:
The change of PELD scores during study | baseline, 3 months, 6 months, 9 months, 12 months
  The PELD score is calculated using the following formula:
  PELD Score = 0.480 * ln (Bilirubin in mg/dL) + 1.857 * ln (INR) - 0.687 * ln (Albumin in g/dL) + 0.436 if the patient is <1 year old + 0.667 if there growth failure
The change of albumin (Liver function) | up to the 12-month period following treatment
  Levels of albumin (g/dL)
The change of total bilirubin (Liver function) | up to the 12-month period following treatment
  Total bilirubin level (mg/dL)
The change of prothrombin time | up to the 12-month period following treatment
  Prothrombin time (second)
The change of liver biopsy | up to the 12-month period following treatment
  change of liver biopsy

SECONDARY OUTCOMES:
The number of Adverse Events (AE) and Serious Adverse Events (SAE) | baseline, 3 months, 6 months, 9 months, 12 months (time frame: up to the 12-month period following treatment)
  Adverse Events (AE) and Serious Adverse Events (SAE) after MSC transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Liem Nguyen, Principal Investigator — Vinmec Research Institute of Stem Cell and Gene Technology
Locations (2):
- Vietnam (2):
  - Vinmec International Hospital Times City, Hanoi, Hanoi
  - Vinmec Research Institute of Stem cell and Gene Technology, Hanoi

IPD SHARING:
Plan to Share IPD: No
When the study complete

REFERENCES:
- [Derived] Nguyen TL, Nguyen HP, Bui TH, Phan TKT, Ngo DM, Ha TTH, Tran TT, Luu NAT, Phan TK, Ho PD. Outcomes of Allogeneic Umbilical Cord Mesenchymal Stem Cell Infusion for Liver Cirrhosis Due to Biliary Atresia After Kasai Operation. J Pediatr Surg. 2025 Nov;60(11):162624. doi: 10.1016/j.jpedsurg.2025.162624. Epub 2025 Sep 2. PMID 40907882